CLINICAL TRIAL: NCT06747286
Title: The Effectiveness of Virtual Game Simulation Method Designed for Patient Safety in Nursing Students
Brief Title: Virtual Game Simulation in Patient Safety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Derya Avan Çınar, Principal Investigator, Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SBU-SBEH-DAC-01
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Nurse's Role
Keywords: Virtual Game Simulation; Nursing Education; Patient Safety

STUDY DESIGN:
Intervention Model Description: Two groups with an experiment control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): Group to be applied virtual game simulation
  Interventions: Other: Virtual Game Simulation
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: Virtual Game Simulation — A virtual computer game that enables participation in a clinical scenario to measure competence.
  Other Names: experimental
  Arms: Experiment group

SUMMARY:
With the development of technology, virtual game simulation is starting to take an important place in nursing education, which has spread to the virtual world. There are studies conducted with this application, but there are no virtual game simulation studies related to patient safety. The planned study aims to measure nursing students' tendencies and attitudes towards medical errors, satisfaction and self-confidence in nursing practices with a virtual game simulation related to patient safety developed by the researcher.

DETAILED DESCRIPTION:
Simulation, also defined as activities that imitate clinical practices and simulation, are applications that provide competency-based clinical experience in a realistic environment that does not carry the risk of the real situation and is of great importance in terms of patient safety. Virtual game simulation, which includes technology and is one of the simulation applications, is a two-dimensional virtual computer game that includes simulated real people and allows students to actively participate in a clinical scenario. While the use of virtual game simulation in nursing education increases students' critical thinking, decision-making and problem-solving skills, it also provides learning by making mistakes and correcting mistakes by increasing individual development. The use of virtual game simulation in nursing education is necessary and important in ensuring and protecting patient safety. Virtual games, whose main purpose is to learn, have the potential to increase student participation, role-play difficult situations, try new reactions or work on creative solutions.

ELIGIBILITY:
Inclusion Criteria:

* Having taken the Fundamentals of Nursing course,
* Being willing and eager to participate in the study,
* Completing the Data Collection Forms completely,
* Not having any communication problems related to vision or hearing,
* Completing all stages of the simulation training process.

Exclusion Criteria:

* Not having received simulation training regarding patient safety.

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Structured Student Information Form | one month
  The structured student information form, developed by the researcher in line with literature knowledge, includes a total of 13 questions on topics such as students' age, gender, etc.
Modified Simulation Effectiveness Tool | one month
  The measurement tool for students' perceptions of the effectiveness of learning in a simulation environment was designed for self-reporting. The measurement tool has 19 items and four sub-dimensions. It is a 3-point Likert-type scale where the items are scored from 1 to 3. Scored as 1 - "Disagree", 2 - "Partially Agree", 3 - "Strongly Agree". The Cronbach Alpha internal consistency coefficient of the measurement tool is 0.93; the Cronbach Alpha coefficients of its sub-dimensions are 0.83, 0.85, 0.91 and 0.90, respectively. The total score is obtained by summing up all sub-dimension scores.
Simulation Design Scale | one month
  The scale consists of 20 items and five subscales: "Goals and Information", "Support", "Problem Solving", "Feedback/Guided Reflection", and "Authenticity". The scale consists of two parts. The first part measures whether the best simulation design elements were applied in the simulation application. This section includes the statements "Strongly Disagree", "Disagree", "Undecided", "Agree", "Strongly Agree", and "Not Appropriate". The second part measures how important the simulation application is for the students. This section includes the statements "Not Important", "Partially Important", "Undecided", "Important", and "Very Important". Cronbach's Alpha values for the subheadings vary between 0.73 and 0.86. The score range is determined as 1 point being the lowest and 5 points being the highest. The scale is scored by dividing the total score given to the answers by the number of items.
Student Satisfaction and Learning Self-Confidence Scale | one month
  It consists of two sub-dimensions, "satisfaction with learning" and "self-confidence", and a total of 13 items. The 13th item in the scale is reverse coded. The answer options are 5= Strongly agree, 4= Agree, 3= Undecided: Neither agree nor disagree, 2= Disagree, 1= Strongly disagree. The score is obtained from the sum of the items in the scale. The highest score that can be obtained from the scale is 65, the lowest score is 13. The internal consistency coefficient of the scale was found to be 0.94.
Medical Error Scale for Nursing Students | one month
  The scale was prepared in a 5-point Likert type consisting of 36 items and 7 sub-dimensions, evaluated as always (5), usually (4), sometimes (3), rarely (2), never (1). The total score range of the scale is between 36 and 180. Scores close to 180 on the scale indicate that student nurses are controlled or careful regarding medical errors, while scores close to 36 indicate that student nurses are not controlled regarding medical errors or may make medical errors.
Attitude Scale on Medical Errors | one month
  The scale consists of 16 items and 3 sub-dimensions. The aim of the scale is to examine the attitudes of healthcare professionals towards medical errors. It has 3 sub-headings: medical error perception (2 items), medical error approach (7 items), and reasons for medical errors (7 items). The scale is a five-point Likert-type scale. The scores of the answers to the items range from (1) I completely disagree to (5) I completely agree. Questions 10 and 13 under the sub-heading of medical error approach are reverse scored. The cut-off point of the scale is determined as 3. In the scale calculation, the total scale score is obtained by dividing the scale item number. In the sub-dimension calculation, the total score of the sub-dimension is divided by the number of items related to the relevant sub-dimension. The obtained score is between 1 and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Derya AVAN ÇINAR, Study Principal Investigator, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Health Sciences University Hamidiye Faculty of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No